CLINICAL TRIAL: NCT02017444
Title: Lowering Intracranial Pressure in Idiopathic Intracranial Hypertension: Assessing the Therapeutic Efficacy and Safety of an 11β-hydroxysteroid Dehydrogenase Type 1 Inhibitor (AZD4017). Phase II Study.
Brief Title: Safety and Effectiveness of 11b-Hydroxysteroid Dehydrogenase Type 1 Inhibitor (AZD4017) to Treat Idiopathic Intracranial Hypertension.
Acronym: IIH:DT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Principal Investigator, Dr Alexandra Sinclair, Chief Investigator, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RG_13-022; 2013-003643-31 (EudraCT Number); MR/K015184/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: Pseudotumor Cerebri; Benign Intracranial Hypertension; Headaches; Tinnitus; Papilledema; Blindness; Optic Disk; Intracranial Hypertension; Clinical Trial, Phase 2; 11beta-Hydroxysteroid Dehydrogenase Type 1; Obesity
MeSH Terms: conditions — Pseudotumor Cerebri; Headache; Tinnitus; Papilledema; Blindness; Intracranial Hypertension; Obesity | interventions — 2-(1-(5-(cyclohexylcarbamoyl)-6-propylsulfanylpyridin-2-yl)-3-piperidyl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matched placebo tablet B.D for 12 weeks
  Interventions: Other: Placebo
- AZD4017 (11b-HSD1 inhibitor) (Active Comparator): AZD4017 400mg tablet B.D. for 12 weeks
  Interventions: Drug: AZD4017

INTERVENTIONS:
Drug: AZD4017
  Other Names: 11b-Hydroxysteroid dehydrogenase type 1 inhibitor
  Arms: AZD4017 (11b-HSD1 inhibitor)
Other: Placebo — Matched placebo (matched to AZD4017 arm)
  Arms: Placebo

SUMMARY:
Assessing the safety and effectiveness of a 11-βhydroxysteroid dehydrogenase type 1 inhibitor (AZD4017), in a placebo controlled trial, in acute idiopathic intracranial hypertension (IIH) IIH is a condition of young, overweight women with characteristic raised intracranial pressure (pressure around the brain) leading to papilloedema (swelling of the nerve supplying the eye), visual loss and headaches. Medical literature (Cochrane review) demonstrates there is little evidence for the treatments used for IIH. Weight control appears the most effective method of improving symptoms but weight loss is difficult to maintain. 11β-hydroxysteroid dehydrogenase type 1 (11β-HSD1) is an enzyme which regulates local steroid levels and our previous research suggests it may influence the production of brain fluid(cerebrospinal fluid or CSF). 11β-HSD1 levels fall with weight loss and this is associated with with decreased intracranial pressure.

Our primary outcome is to determine whether AZD4017, an inhibitor of 11β-HSD1, will reduce the pressure in the brain and as a consequence improve IIH. Patients are eligible to enter the study if they are between 18-55 years old with acute (<6 months) IIH, signs of active disease (papilloedema and raised CSF pressure (>25 cmH20)), no other major illnesses and have no plans for pregnancy during the study period.

This is an MRC funded single centre, phase II, double-blinded, randomised control drug trial. It will be conducted at the University Hospital Birmingham and the University of Birmingham will act as Sponsor. Eligible participants will be randomly assigned to AZD4017 or a placebo ('dummy' with no active drug) for 3 months with a follow up a month later. Investigations during the study will include bloods, urine samples, pregnancy tests, lumbar punctures, DXA scans and small fat/skin biopsies. Participants will benefit from increased monitoring and a potential improvement in their condition.

We hypothesise that specific inhibition of 11β-HSD1 will decrease intracranial pressure and consequently treat patients with IIH, thus opening a new and entirely novel therapeutic avenue.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Female patients between 18 and 55 years
* Diagnosis of IIH by the Modified Dandy criteria1 with:

  1. acute (<6 months),
  2. active disease (papilloedema (Frisen grade greater than or equal to 1),
  3. significantly raised ICP > 25cmH2O)
  4. normal brain imaging during previous routine diagnostic work up (evaluated by either magnetic resonance venography or computerised tomography with venography).
* Patients must be willing to use one form of highly effective non-hormonal contraception. This would include:

  1. a vasectomised partner (sole partner) or tubal occlusion or
  2. copper containing IUD - all of which should be used in addition to a diaphragm or cervical/vault caps with barrier contraceptive (condom or spermicidal foam/gel/film/suppository)
  3. true abstinence (when this is in line with the preferred and usual lifestyle of the subject. Women should have been stable on their chosen method of birth control for a minimum of 2 months before entering the trial. Patients must agree to undergo a β-hCG pregnancy test and urine dipstick test at screening and urine dipstick testing at all trial visits (including the final follow up visit 4 weeks after discontinuation of study treatment). Note: the use of contraception and pregnancy testing would not be required if the screening LH/FSH levels demonstrate the patient is post-menopausal.
* Participants are able to continue other medications to treat their IIH e.g. acetazolamide, diuretics but this dose must remain fixed throughout the study.
* Patients who take aspirin therapy will be asked to discontinue aspirin 3 days prior to fat and skin biopsy if clinically safe to do so.
* Placebo treatment for the duration of the study must not be considered detrimental to the patient.
* Must be able to understand the consent form and comply with study requirements.

Exclusion Criteria:

* Optic nerve sheath fenestration.
* Patients who undergo CSF shunt insertion (which is not elective or pre- planned) during the study, as a result of deterioration will be withdrawn from the study.
* Abnormal neurological examination (aside from papilloedema and consequent visual loss or VI nerve palsy).
* Subjects with a secondary cause of raised intracranial pressure will be excluded (venous thrombosis, anaemia, drug causes (lithium, vitamin A, tetracycline or others deems responsible for the condition).
* Abnormal CSF contents (except for that compatible with a traumatic LP).
* Unable to perform a visual field reliably.

General Exclusion Criteria:

* Positive hCG or urine dipstick pregnancy test or planning to conceive in the 4 study months.
* Have eGFR calculated by MDRD equation of <60ml/min/1.73m2.
* Have any endocrine disorder, e.g. thyroid dysfunction. This excludes PCOS where there is a known association to IIH.
* Suspicion of or known Gilbert's disease.
* CK >2 x ULN on 2 consecutive measurements.
* ALT and/or AST >2 x ULN.
* ALP > ULN.
* Bilirubin (total) > 2 x ULN.
* Must not have donated blood within 2 months of screening and avoid further donations for 4 months following the study.
* Patient is, at the time of signing the informed consent, a user of recreational or illicit drugs (including marijuana) or has had a recent history (within the last year) of drug or alcohol abuse or dependence.
* Pregnant or breastfeeding mothers, unless willing to discontinue breastfeeding by the baseline visit.
* Have uncontrolled systemic hypertension (BP >160/90), on 3 successive measurements on the morning of the screening visit.
* Are receiving systemic (including vaginal/rectal) glucocorticoid treatment at the time of the screening visit. Note: Topical and inhaled are acceptable
* Are taking any hormone-based medication, including hormone contraceptives, at the time of screening.
* Are taking probenecid at the time of the screening visit.
* Have any screening laboratory abnormality that, in the investigator's judgement, is considered to be clinically significant or any screening laboratory value which is outside the Sponsor specified ranges at screening; testing may be repeated but must be resolved prior to the baseline visit.
* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation or will influence the results .
* History or presence of significant gastrointestinal, hepatic , or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IP as judged by the investigator.
* Have been involved in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Have participated in any other interventional study within 1 month prior to the screening visit. Participation in the IIH National database or other observational studies will not prevent enrolment to this study.
* Previous randomisation for treatment in the present study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-04-25 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sinclair, MbChb PhD, Principal Investigator — University of Birmingham
Locations (1):
- University Hospital Birmingham (Queen Elizabeth Hospital), Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gomez C, Alimajstorovic Z, Othonos N, Winter DV, White S, Lavery GG, Tomlinson JW, Sinclair AJ, Odermatt A. Identification of a human blood biomarker of pharmacological 11beta-hydroxysteroid dehydrogenase 1 inhibition. Br J Pharmacol. 2024 Mar;181(5):698-711. doi: 10.1111/bph.16251. Epub 2023 Oct 19. PMID 37740611
- [Derived] Grech O, Seneviratne SY, Alimajstorovic Z, Yiangou A, Mitchell JL, Smith TB, Mollan SP, Lavery GG, Ludwig C, Sinclair AJ. Nuclear Magnetic Resonance Spectroscopy Metabolomics in Idiopathic Intracranial Hypertension to Identify Markers of Disease and Headache. Neurology. 2022 Oct 17;99(16):e1702-e1714. doi: 10.1212/WNL.0000000000201007. PMID 36240084
- [Derived] Hardy RS, Botfield H, Markey K, Mitchell JL, Alimajstorovic Z, Westgate CSJ, Sagmeister M, Fairclough RJ, Ottridge RS, Yiangou A, Storbeck KH, Taylor AE, Gilligan LC, Arlt W, Stewart PM, Tomlinson JW, Mollan SP, Lavery GG, Sinclair AJ. 11betaHSD1 Inhibition with AZD4017 Improves Lipid Profiles and Lean Muscle Mass in Idiopathic Intracranial Hypertension. J Clin Endocrinol Metab. 2021 Jan 1;106(1):174-187. doi: 10.1210/clinem/dgaa766. PMID 33098644
- [Derived] Markey KA, Ottridge R, Mitchell JL, Rick C, Woolley R, Ives N, Nightingale P, Sinclair AJ. Assessing the Efficacy and Safety of an 11beta-Hydroxysteroid Dehydrogenase Type 1 Inhibitor (AZD4017) in the Idiopathic Intracranial Hypertension Drug Trial, IIH:DT: Clinical Methods and Design for a Phase II Randomized Controlled Trial. JMIR Res Protoc. 2017 Sep 18;6(9):e181. doi: 10.2196/resprot.7806. PMID 28923789

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD4017 (11b-HSD1 Inhibitor): AZD4017 400mg tablet B.D. for 12 weeks
  AZD4017
Period: Overall Study
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Started | 14 | 17
Completed | 12 | 17 (NB: One participant did not complete primary outcome.)
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Patient withdrawn day after randomisation as found to be ineligible. Did not return for follow up. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor) | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (8) | 30.1 (5.9) | 31.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 13 | 16 | 29
  Asian/Asian British - Pakistani | 0 | 1 | 1
  Asian/Asian British - Other Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14 | 17 | 31
Taking acetazolamide (yes/no) [Count of Participants; unit: Participants]
  Yes | 4 | 6 | 10
  No | 10 | 11 | 21
Opening LP pressure (cmCSF) [Mean (Standard Deviation); unit: cmCSF] | 32.7 (4.8) | 33.7 (6.3) | 33.3 (5.6)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 108 (42.3) | 97.9 (21.3) | 102.6 (32.3)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 41.2 (16.6) | 37.3 (7.2) | 39.2 (12.6)
Headache Impact Test 6 (HIT-6) Score [Mean (Standard Deviation); unit: HIT-6 score (higher is worse)] | 63.4 (8.1) | 63.8 (8.2) | 63.6 (8)
Frisen grading (Worst eye) [Count of Participants; unit: Participants] — Papilloedema were evaluated at the end of trial follow up using stereoscopic fundus photographs by masked neuro-ophthalmologists to grade the images according to Frisen classification. There are 6 grades, 0-5, 5 being the worst.
  The modified Frisén scale for grading papilledema is as follows:
  Grade 1 - C-Shaped halo with a temporal gap
  Grade 2 - The halo becomes circumferential
  Grade 3 - Loss of major vessels as they leave the disc
  Grade 4 - Loss of major vessels on the disc
  Grade 5 - Grade IV + partial or total obscuration of all vessels on the disc
  Participants
    1 | 2 | 4 | 6
    2 | 5 | 9 | 14
    3 | 3 | 0 | 3
    4 | 1 | 2 | 3
    5 | 0 | 1 | 1
    missing | 1 | 0 | 1
Presence of Pulsatile Tinnitus [Count of Participants; unit: Participants]
  Presence | 13 | 12 | 25
  Absence | 1 | 5 | 6
Presence of visual loss [Count of Participants; unit: Participants]
  Presence | 8 | 4 | 12
  Absence | 6 | 13 | 19
Presence of diplopia [Count of Participants; unit: Participants]
  Presence | 5 | 7 | 12
  Absence | 9 | 10 | 19
Presence of Visual obscuration [Count of Participants; unit: Participants]
  Presence | 6 | 6 | 12
  Absence | 8 | 11 | 19
Presence of headache [Count of Participants; unit: Participants]
  Presence | 14 | 16 | 30
  Absence | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Pressure
Description: ICP measured by lumbar puncture in cmCSF as the change from week 0 and week 12 of treatment, measured at baseline and week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cmCSF
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 12 | 16
cmCSF | -0.3 (5.9) | -4.3 (5.7)

2. Secondary Outcome: Tinnitus
Description: The temporal change in IIH symptoms (presence or absence of tinnitus), measured at baseline and week 12
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 12 | 17
Participants
  Presence | 7 | 9
  Absence | 5 | 8

3. Secondary Outcome: Anthropometric Measurements (BMI)
Description: The temporal change in Body Mass Index (in kg/m^2) over 12 weeks of treatment, measured at baseline and week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 11 | 17
kg/m^2 | 37.4 (8.4) | 37.5 (6.9)

4. Secondary Outcome: Visual Loss
Description: The temporal change in IIH symptoms (presence or absence of visual loss, measured at baseline and week 12
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 11 | 17
Participants
  Presence | 7 | 6
  Absence | 4 | 11

5. Secondary Outcome: Diplopia
Description: The temporal change in IIH symptoms (presence or absence of diplopia, measured at baseline and week 12
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 12 | 17
Participants
  Presence | 1 | 2
  Absence | 11 | 15

6. Secondary Outcome: Visual Obscuration
Description: The temporal change in IIH symptoms (presence or absence of visual obscuration, measured at baseline and week 12
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 11 | 17
Participants
  Presence | 2 | 2
  Absence | 9 | 15

7. Secondary Outcome: Headache
Description: The temporal change in IIH symptoms (presence or absence of headache, measured at baseline and week 12
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 12 | 17
Participants
  Presence | 10 | 13
  Absence | 2 | 4

8. Secondary Outcome: Visual Acuity
Description: The temporal change in IIH visual function in both eyes (measured by LogMAR (log of the minimum angle of resolution) chart to assess visual acuity, between the baseline to week 12, measured at baseline and week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: LogMAR (log of the minimum angle of reso
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 14 | 17
LogMAR (log of the minimum angle of reso
  Baseline LVA worst eye | 0.13 (0.22) | 0.08 (0.23)
  Week 12 LVA worst eye | 0.09 (0.18) | 0.06 (0.15)

9. Secondary Outcome: Papilloedema
Description: The temporal change in papilloedema (evaluated at the end of trial follow up using stereoscopic fundus photographs by masked neuro-ophthalmologists to grade the images according to Frisen classification) measured at baseline and week 12. There are 6 grades, 0-5, 5 being the worst.
  The modified Frisén scale for grading papilledema using fundus photography is as follows:
  Grade 1 - C-Shaped halo with a temporal gap
  Grade 2 - The halo becomes circumferential
  Grade 3 - Loss of major vessels as they leave the disc
  Grade 4 - Loss of major vessels on the disc
  Grade 5 - Criteria of Grade IV + partial or total obscuration of all vessels on the disc
  For further details see e.g. Scott, C.J., et al., Diagnosis and grading of papilledema in patients with raised intracranial pressure using optical coherence tomography vs clinical expert assessment using a clinical staging scale. Arch. Ophthalmol, 2010. 128(6): p. 705-711.
Time Frame: 12 weeks
Population: NB: assessment missed for one participant at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 12 | 16
Participants
  Frisen grade 0 baseline: number analyzed (Participants) | 11 | 16
  Frisen grade 0 baseline | 0 | 0
  Frisen grade 0 week 12 | 0 | 2
  Frisen grade 1 baseline: number analyzed (Participants) | 11 | 16
  Frisen grade 1 baseline | 2 | 4
  Frisen grade 1 week 12 | 2 | 5
  Frisen grade 2 baseline: number analyzed (Participants) | 11 | 16
  Frisen grade 2 baseline | 5 | 9
  Frisen grade 2 week 12 | 6 | 8
  Frisen grade 3 baseline: number analyzed (Participants) | 11 | 16
  Frisen grade 3 baseline | 3 | 0
  Frisen grade 3 week 12 | 3 | 0
  Frisen grade 4 baseline: number analyzed (Participants) | 11 | 16
  Frisen grade 4 baseline | 1 | 2
  Frisen grade 4 week 12 | 1 | 1
  Frisen grade 5 baseline: number analyzed (Participants) | 11 | 16
  Frisen grade 5 baseline | 0 | 1
  Frisen grade 5 week 12 | 0 | 0

10. Secondary Outcome: Headache-associated Disability
Description: The change in headache associated disability through the headache impact test-6 score (HIT 6), measured at baseline and week 12. This is scored 11-66 with higher scores indicating worse headache.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score on HIT-6 scale
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 11 | 15
Score on HIT-6 scale | 59.8 (7.9) | 60.1 (11.6)

11. Secondary Outcome: Adverse Events
Description: The safety and tolerability profile of AZD4017 in female patients with IIH through adverse event reporting and safety bloods.
Time Frame: 16 weeks
Measure: Number; unit: AEs related to intervention
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 14 | 17
AEs related to intervention | 0 | 9

12. Secondary Outcome: Serious Adverse Events
Description: as for outcome 11
Time Frame: 16 weeks
Measure: Number; unit: Serious adverse events
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 14 | 17
Serious adverse events | 1 | 0

13. Secondary Outcome: OCT Total Average Retinal Nerve Fibre Layer Thickness (μm)
Description: The temporal change in OCT Total average retinal nerve fibre layer thickness (μm), measured at baseline and week 12
Time Frame: 12 weeks
Population: NB: assessment missed in participants of both arms due to centre capacity.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 14 | 17
μm
  Total average retinal nerve fibre layer baseline worst ete | 158.4 (83) | 152 (68.7)
  Total average retinal nerve fibre layer week 12 worst eye: number analyzed (Participants) | 11 | 15
  Total average retinal nerve fibre layer week 12 worst eye | 143.2 (78.7) | 139.7 (56.3)

14. Secondary Outcome: Visual Field Mean Deviation
Description: The temporal change in IIH visual function in both eyes using automated perimetry (Humphrey 24-2 central threshold) to measure the visual field mean deviation between the baseline to week 12
Time Frame: 12 weeks
Population: NB: assessment at 12 weeks not completed for 2 participants.
Measure: Mean (Standard Deviation); unit: Visual field mean deviation
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 14 | 17
Visual field mean deviation
  Baseline MD worst eye | -3.4 (6.8) | -6.1 (5.4)
  Week 12 MD worst eye: number analyzed (Participants) | 12 | 17
  Week 12 MD worst eye | -2.2 (3.1) | -3.4 (3.2)

15. Secondary Outcome: Log Contrast Sensitivity
Description: The temporal change in IIH visual function in both eyes using a Pelli-Robson chart to evaluate log contrast sensitivity between the baseline to week 12
Time Frame: 12 weeks
Population: NB: assessment at 12 weeks not completed for 2 participants (placebo).
Measure: Mean (Standard Deviation); unit: Log contrast senstivity
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
Number analyzed (Participants) | 12 | 13
Log contrast senstivity
  Baseline LCS worst eye | 1.63 (0.16) | 1.63 (0.22)
  Week 12 LCS worst eye: number analyzed (Participants) | 10 | 13
  Week 12 LCS worst eye | 1.66 (0.12) | 1.65 (0.15)

ADVERSE EVENTS:
Arm/Group | Placebo | AZD4017 (11b-HSD1 Inhibitor)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/17
Other Adverse Events (participants affected / at risk) | 11/14 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | AZD4017 (11b-HSD1 Inhibitor) (N=17)
IIH exacerbation (Eye disorders) | 1 (1) | 0 (0) — IIH exacerbation requiring acute intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | AZD4017 (11b-HSD1 Inhibitor) (N=17)
Cardiovascular (Cardiac disorders) | 1 | 1
Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Gastro-intestinal (Gastrointestinal disorders) | 3 | 8
Genito-urinary (General disorders) | 0 | 6
Endocrine (Endocrine disorders) | 1 | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 | 6
Neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neurological (Nervous system disorders) | 3 | 7
Psychological (Psychiatric disorders) | 4 | 4
Immunological (Immune system disorders) | 1 | 0
Dermatological (General disorders) | 5 | 2
Allergies (General disorders) | 0 | 1
Eyes, ear, nose, throat (Ear and labyrinth disorders) | 6 | 12
Other (General disorders) | 5 | 7 — tiredness; hot sweats; flu like symptoms; disrupted sleep; toothache/infection; breast pain; menstrual problems for more than 3 weeks; mouth ulcers; a cold; transient nausea and height headaches

LIMITATIONS AND CAVEATS:
A duration of 12 weeks was chosen for the evaluation of safety and tolerability, being the longest duration of dosing to date with AZD4017. This may not have been enough for meaningful evaluation of clinical outcomes.

The sample size is small, which may have reduced power and limited meaningful evaluation of clinical measures: the trial was not designed to establish significant changes in the secondary clinical outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No